CLINICAL TRIAL: NCT00389792
Title: A Randomized, Double-Blind, Placebo-Controlled Study of ATI-2042 in Patients With Paroxysmal Atrial Fibrillation and Pacemakers With Atrial Fibrillation Data Logging Capabilities
Brief Title: Efficacy and Safety Study of an Antiarrhythmic Drug to Treat Atrial Fibrillation in Patients With Pacemakers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARYx Therapeutics (Industry)
Responsible Party: Eppie Chang, Senior Director of Clinical Operations, ARYx Therapeutics, 6300 Dumbarton Circle, Fremont, CA 94555
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATI 2042-CLN 205
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — celivarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ATI-2042 200 mg (No Intervention)
  Interventions: Drug: ATI-2042; Drug: ATI-2042 200 mg
- ATI-2042 400 mg (No Intervention)
  Interventions: Drug: ATI-2042; Drug: ATI-2042 200 mg
- ATI-2042 600 mg (No Intervention)
  Interventions: Drug: ATI-2042; Drug: ATI-2042 200 mg
- ATI-2042 Placebo (No Intervention)
  Interventions: Drug: ATI-2042; Drug: ATI-2042 200 mg

INTERVENTIONS:
Drug: ATI-2042 — no intervention
Drug: ATI-2042 200 mg — To stop the dosing of ATI-2042 for a designated time frame as determined by the medical monitor and Principal Investigator.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an investigational antiarrhythmic drug (ATI-2042) in the treatment of atrial fibrillation in patients with a dual chamber pacemaker.

DETAILED DESCRIPTION:
ATI-2042 is being developed as an alternative to amiodarone, which is considered a first-line therapy for patients with atrial fibrillation and is known to have serious side effects. ATI-2042 was designed to have a reduced plasma half-life and a lower volume of distribution, which is expected to result in an improved safety profile. In contrast to amiodarone, ATI-2042 undergoes rapid metabolism via plasma and tissue esterases, which may reduce tissue accumulation and toxicity. The current trial will determine if ATI-2042 retains the efficacy profile of amiodarone without the side effects attributable to tissue accumulation seen with long-term dosing.

This study is an early phase trial and some specific protocol information is proprietary and not publicly available at this time. (Full information is available to trial participants.)

ELIGIBILITY:
Inclusion Criteria:

* Proven paroxysmal atrial fibrillation
* Pacemaker with appropriate AF diagnostics and recording capabilities

Exclusion Criteria:

* Known allergy to Amiodarone or previous treatment for severe Amiodarone toxicity
* Cardioversion within one month of screening
* Severe left ventricular dysfunction or CHF with NYHA Class III or above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Efficacy Measure: Atrial Fibrillation Burden
Safety Measures: ECG, Laboratory and Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ezekowitz, MBChB, PhD, Study Chair — Main Line Health; Olga Bandman, MD, Study Director — ARYx Therapeutics
Locations (38):
- United States (27):
  - ARYx Investigational Site, Phoenix, Arizona
  - ARYx Investigational Site, Scottsdale, Arizona
  - ARYx Investigational Site, Tucson, Arizona
  - ARYx Investigational Site, Larkspur, California
  - ARYx Investigational Site, Aurora, Colorado
  - ARYx Investigational Site, Hollywood, Florida
  - ARYx Investigational Site, Jacksonville Beach, Florida
  - ARYx Investigational Site, Atlanta, Georgia
  - ARYx Investigational Site, Marietta, Georgia
  - ARYx Investigational Site, Chicago, Illinois
  - ARYx Investigational Site, Towson, Maryland
  - ARYx Investigational Site, Saginaw, Michigan
  - ARYx Investigational Site, Minneapolis, Minnesota
  - ARYx Investigational Site, St Louis, Missouri
  - ARYx Investigational Site, Lincoln, Nebraska
  - ARYx Investigational Site, Warren Township, New Jersey
  - ARYx Investigational Site, Albuquerque, New Mexico
  - ARYx Investigational Site, Buffalo, New York
  - ARYx Investigational Site, Hershey, Pennsylvania
  - ARYx Investigational Site, Wynnewood, Pennsylvania
  - ARYx Investigational Site, Charleston, South Carolina
  - ARYx Investigational Site, Nashville, Tennessee
  - ARYx Investigational Site, Austin, Texas
  - ARYx Investigational Site, Houston, Texas
  - ARYx Investigational Site, Burlington, Vermont
  - ARYx Investigational Site, Newport News, Virginia
  - ARYx Investigational Site, Charleston, West Virginia
- Canada (11):
  - ARYx Investigational Site, Edmonton, Alberta
  - ARYx Investigational Site, Campbell River, British Columbia
  - ARYx Investigational Site, Vancouver, British Columbia
  - ARYx Investigational Site, Victoria, British Columbia
  - ARYx Investigational Site, London, Ontario
  - ARYx Investigational Site, Niagara Falls, Ontario
  - ARYx Investigational Site, Ottawa, Ontario
  - ARYx Investigational Site, Montreal, Quebec
  - ARYx Investigational Sites, Montreal, Quebec
  - ARYx Investigational Site, Sherbrooke, Quebec
  - ARYx Investigational Site, Terrebonne, Quebec